CLINICAL TRIAL: NCT01523405
Title: A Non-Interventional Study To Evaluate Diabetes Related Quality Of Life, Frequency And Impact Of Hypoglycemia In Type 2 Diabetes Patients On Pharmacotherapy (INSIGHT)
Brief Title: A Non-Interventional Study To Evaluate Diabetes Related Quality Of Life, Frequency And Impact Of Hypoglycemia In T2DM
Acronym: INSIGHT
Status: Completed | Type: Observational
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Other Study IDs: NIS-CIN-XXX-2011/3
Record Dates: First submitted 2012-01-30; First posted 2012-02-01 (Estimated); Last update posted 2014-09-08 (Estimated); Status verified 2014-09

CONDITIONS: Type II Diabetes Mellitus
Keywords: Non Interventional Study, Type II Diabetes Mellitus, Quality of Life
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- 1

SUMMARY:
This is a non-interventional, cross sectional, multicentric study in T2DM patients which will involve a single visit for study related procedures. This study will be conducted in approximately 5,000 patients at around 300 hospitals/primary care clinics across India. Approximately 18-20 patients per site will be enrolled. This study has been designed to evaluate diabetes related quality of life (DQoL), frequency and impact of hypoglycaemia in relation to HbA1c control and to assess disease modifying variables-BMI and BP in T2DM patients on oral / injectable anti-diabetic drugs with/without insulin therapy.

DETAILED DESCRIPTION:
A Non-Interventional Study To Evaluate Diabetes Related Quality Of Life, Frequency And Impact Of Hypoglycemia In Type 2 Diabetes Patients On Pharmacotherapy (INSIGHT)

ELIGIBILITY:
Inclusion Criteria:

* Patients with diagnosis of T2DM for > 1 year prior to entry in the study willing and able to complete the questionnaire and on pharmacotherapy
* Patients who are currently treated with a single or combination of injectable/oral antidiabetic drugs with or without insulin therapy
* Treatment type must be unchanged in the previous 3 months. However, dose modifications are allowed
* Patients who agree to participate in the study and give their written informed consent

Exclusion Criteria:

* Patients with type 1 diabetes
* Patients with diabetic ketoacidosis and/or hyperosmolar hyperglycaemic state
* Patients with secondary diabetes (including disease of the exocrine pancreas, endocrinopathies)
* Patients with concurrent treatment involving systemic glucocorticoids. However, inhaled, locally injected and topical use of glucocorticoids is allowed
* Patients suffering from severe cardiac, hepatic, renal diseases as judged by the investigator
* Any condition of the patient which may have an impact on objective and outcome of the trial example: patients currently undergoing major/ minor surgical

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Approximately 5,000 adult patients (≥ 18 years) diagnosed with T2DM will be randomly selected from around 300 hospitals/primary care clinics across India to participate in this study.
Sampling Method: Non-Probability Sample
Enrollment: 4911 (Actual)
Dates: Start 2012-03; Primary Completion 2013-02 (Actual); Study Completion 2013-02 (Actual)

PRIMARY OUTCOMES:
Diabetic Quality of Life using Modified 15 item DQoL (MDQoL) questionnaire | 2nd February 2012 - 2nd August 2012

SECONDARY OUTCOMES:
HbA1c and its correlation with frequency of hypoglycemia | 2nd February 2012 - 2nd August 2012
Frequency and impact of hypoglycemia using HFS-II (worry subscale) | 2nd February 2012 - 2nd August 2012
Disease modifying variables Body Mass Index (BMI) and Blood Pressure (BP) | 2nd February 2012 - 2nd August 2012

CONTACTS AND LOCATIONS:
Overall Officials: Abhay Raut, MD, Principal Investigator — Prashanti Clinic,; Sashi Kumar, MBBS, Principal Investigator — Dianova Diabetes Centre; Subodh Chandra, MD, Principal Investigator — Chandra Medicals Pvt. Ltd; Debashish Maji, MD, DM, Principal Investigator — Calcutta Diabetes and endocrine Foundation,; Mayur Patel, MD, Principal Investigator — Swasthya (All India Institute of Diabetes and Research); Nallaperumal Sivagnam, MBBS, Principal Investigator — Swamy Diabetes Centre,
Locations (70):
- India (70):
  - Research Site, Vijayawada, Andhara Pradesh
  - Research Site, Hanamkoda, Andhra Pradesh
  - Research Site, Hyderabad, Andhra Pradesh
  - Research Site, Kammam, Andhra Pradesh
  - Research Site, Khammam, Andhra Pradesh
  - Research Site, Kurnool, Andhra Pradesh
  - Research Site, Nellore, Andhra Pradesh
  - Research Site, Vijayawada, Andhra Pradesh
  - Research Site, Visakhapatnam, Andhra Pradesh
  - Research Site, Guwahati, Assam
  - Research Site, Mysore, Bangalore
  - Research Site, Bilāspur, Chhattisgarh
  - Research Site, Raipur, Chhattisgarh
  - Research Site, Mapusa, Goa
  - Research Site, Ahemdabad, Gujarat
  - Research Site, Ahmedabad, Gujarat
  - Research Site, Anand, Gujarat
  - Research Site, Chennai, Gujarat
  - Research Site, Nadiād, Gujarat
  - Research Site, Vadodara, Gujarat
  - Research Site, Karnāl, Haryana
  - Research Site, Panchkula, Haryana
  - Research Site, Dhanbad, Jharkhand
  - Research Site, Ranchi, Jharkhand
  - Research Site, Bangalore, Karnataka
  - Research Site, Kanpur, Karnataka
  - Research Site, Mangalore, Karnataka
  - Research Site, Mysore, Karnataka
  - Research Site, Trichy, Karnataka
  - Research Site, Hubli, Karnatka
  - Research Site, Mangalore, Karnatka
  - Research Site, Mysore, Karnatka
  - Research Site, Kannur, Kerala
  - Research Site, Bhopal, Madhya Pradesh
  - Research Site, Gwalior, Madhya Pradesh
  - Research Site, Indore, Madhya Pradesh
  - Research Site, Indore(MP), Madhya Pradesh
  - Research Site, Ujjain, Madhya Pradesh
  - Research Site, Mumbai, Maharashtra
  - Research Site, Pune, Maharashtra
  - Research Site, Pune, Mahrastra
  - Research Site, Delhi, National Capital Territory of Delhi
  - Research Site, Delhi, New Delhi
  - Research Site, New Delhi, New Delhi
  - Research Site, New Delh, New Delhi
  - Research Site, Bhubaneswar, Odisha
  - Research Site, Puducherry, Puducherry
  - Research Site, Ludhiana, Punjab
  - Research Site, Jaipur, Rajasthan
  - Research Site, Jodhpur, Rajasthan
  - Research Site, Kota, Rajasthan
  - Research Site, Pushkar, Rajasthan
  - Research Site, Chennai, Tamil Nadu
  - Research Site, Coimbatore, Tamil Nadu
  - Research Site, Cuddlore, Tamil Nadu
  - Research Site, Kanchipuram, Tamil Nadu
  - Research Site, Karaikal, Tamil Nadu
  - Research Site, Madurai, Tamil Nadu
  - Research Site, Thuckalay, Tamil Nadu
  - Research Site, Trichy, Tamil Nadu
  - Research Site, Vellore, Tamil Nadu
  - Research Site, Bhilāi, Uttar Pradesh
  - Research Site, Fatepur, Uttar Pradesh
  - Research Site, Ghaziabad, Uttar Pradesh
  - Research Site, Gorakhpur, Uttar Pradesh
  - Research Site, Kanpur, Uttar Pradesh
  - Research Site, Lucknow, Uttar Pradesh
  - Research Site, Noida, Uttar Pradesh
  - Research Site, Kolkata, West Bangal
  - Research Site, Kolkata, West Bengal